CLINICAL TRIAL: NCT06444009
Title: Neoadjuvant Immunotherapy in Combination With Chemotherapy in Resectable Head and Neck Cancer：A Randomized, Phase II Study
Brief Title: A Phase II Study of Neoadjuvant Immunotherapy in Combination With Chemotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Liu (Other)
Responsible Party: Sponsor-Investigator, Lei Liu, professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-C-W-0001
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Locally advanced head and neck squamous cell carcinoma; Neoadjuvant therapy; Immunotherapy; AK112
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Inosine Triphosphate; Cytidine Triphosphate

STUDY DESIGN:
Intervention Model Description: A Randomized, Controlled, Phase II Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ivonescimab in combination with Nab-paclitaxel + Cisplatin (Experimental): Neoadjuvant:
  Patients receive ivonescimab in combination with nab-paclitaxel + cisplatin for 3 cycles before surgery.
  Surgery:
  Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Adjuvant:
  pCR: Patients receive adjuvant ivonescimab for 16 cycles.
  no pCR:
  Low/ Medium Risk:
  Patients will be treated with intensity modulation radiation therapy (IMRT) alone. Once radiotherapy is complete these patients will receive adjuvant ivonescimab for 16 cycles
  High Risk:
  All patients will be treated with IMRT concurrent with cisplatin or other standard of care chemoradiotherapy regimen. Once chemoradiotherapy is complete these patients will receive adjuvant ivonescimab for 16 cycles.
  Interventions: Drug: Ivonescimab combined with TP
- Cadonilimab in combination with Nab-paclitaxel + Cisplatin (Experimental): Neoadjuvant:
  Patients receive cadonilimab in combination with nab-paclitaxel + cisplatin for 3 cycles before surgery.
  Surgery:
  Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Adjuvant:
  pCR: Patients receive adjuvant cadonilimab for 16 cycles.
  no pCR:
  Low/ Medium Risk:
  Patients will be treated with intensity modulation radiation therapy (IMRT) alone. Once radiotherapy is complete these patients will receive adjuvant cadonilimab for 16 cycles
  High Risk:
  All patients will be treated with IMRT concurrent with cisplatin or other standard of care chemoradiotherapy regimen. Once chemoradiotherapy is complete these patients will receive adjuvant cadonilimab for 16 cycles.
  Interventions: Drug: Cadonilimab combined with TP
- Penpulimab in combination with Nab-paclitaxel + Cisplatin (Experimental): Neoadjuvant:
  Patients receive penpulimab in combination with nab-paclitaxel + cisplatin for 3 cycles before surgery.
  Surgery:
  Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Adjuvant:
  pCR: Patients receive adjuvant penpulimab for 16 cycles.
  no pCR:
  Low/ Medium Risk:
  Patients will be treated with intensity modulation radiation therapy (IMRT) alone. Once radiotherapy is complete these patients will receive adjuvant penpulimab for 16 cycles
  High Risk:
  All patients will be treated with IMRT concurrent with cisplatin or other standard of care chemoradiotherapy regimen. Once chemoradiotherapy is complete these patients will receive adjuvant penpulimab for 16 cycles.
  Interventions: Drug: Penpulimab combined with TP

INTERVENTIONS:
Drug: Ivonescimab combined with TP — Both interventions all drugs intravenous infusion, D1, once every 3 weeks, a total of 3 cycles.
  Other Names: ITP
  Arms: Ivonescimab in combination with Nab-paclitaxel + Cisplatin
Drug: Cadonilimab combined with TP — Both interventions all drugs intravenous infusion, D1, once every 3 weeks, a total of 3 cycles.
  Other Names: CTP
  Arms: Cadonilimab in combination with Nab-paclitaxel + Cisplatin
Drug: Penpulimab combined with TP — Both interventions all drugs intravenous infusion, D1, once every 3 weeks, a total of 3 cycles.
  Other Names: PTP
  Arms: Penpulimab in combination with Nab-paclitaxel + Cisplatin

SUMMARY:
A Randomized, Phase II Study of ivonescimab or cadonilimab or penpulimab in Combination With Cisplatin and Nab-paclitaxel in Patients With locally advanced head and neck squamous cell carcinoma (HNSCC) eligible for resection.

This proposed study will evaluate the efficacy and safety of preoperative administration of ivonescimab or cadonilimab or penpulimab combined with chemotherapy in HNSCC who are eligible for resection.

DETAILED DESCRIPTION:
In this study, eligible patients will be randomized in a 1:1:1 ratio to either the ivonescimab combined with chemotherapy treatment group (Cohort 1), or the cadonilimab combined with chemotherapy treatment group (Cohort 2), or the penpulimab combined with chemotherapy treatment group (Cohort 3). Pathological response rate will be the primary outcome measures. Adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females； Age：18 to 75 years.
2. Histologically or cytologically confirmed head and neck squamous cell carcinoma (HNSCC).
3. Patients with resectable locally advanced head and neck squamous cell carcinoma (LA-HNSCC).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. No prior treatment for the cancer.
6. Intention to undergo curative treatment.
7. Patients with normal organ function and suitable for immunotherapy combined with chemotherapy and surgery:

   Adequate hematologic function (total white blood cell count ≥ 3.0×10^9/L, absolute lymphocyte count ≥ 0.8×10^9/L, absolute neutrophil count ≥ 1.5×10^9/L, platelets ≥ 100×10^9/L, hemoglobin ≥ 90g/L); Adequate hepatic function (bilirubin level ≤ 2 times the upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN); Adequate renal function (serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula), urine protein <2+ on dipstick or <1g in a 24-hour urine collection); Good cardiac function, i.e., normal or clinically insignificant abnormalities on electrocardiogram (ECG), echocardiogram showing a left ventricular ejection fraction (LVEF) ≥50%; Adequate coagulation function: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN; participants on anticoagulation treatment are eligible if the PT is within the therapeutic range of the anticoagulant;
8. Blood pressure well controlled (defined as systolic blood pressure ≤ 150 mmHg and diastolic blood pressure ≤ 90 mmHg) with or without antihypertensive medication, and no change in antihypertensive treatment within 1 week before the first dose of study medication.
9. Patients with HBV infection capable of having detectable HBV DNA levels (≥10IU/mL or above the limit of quantitation) (manifested as positive for hepatitis B surface antigen (HbsAg) and/or hepatitis B core antibody (anti-HBc)) must receive antiviral therapy according to clinical practice at the site before randomization to ensure adequate viral suppression. Patients must maintain antiviral therapy during the study and for 6 months after the last dose of study treatment. Patients who are anti-HBc positive but do not have detectable HBV DNA (<10IU/mL or below the limit of quantitation) are not required to receive antiviral therapy unless their HBV DNA levels exceed 10IU/mL or the limit of quantitation during treatment.
10. Women of childbearing potential (15-49 years old) must have a negative pregnancy test within 7 days before starting treatment; patients of childbearing potential must agree to use effective contraception to ensure they do not become pregnant during the study period and for 3 months after stopping treatment.
11. Participants voluntarily join the study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Patients who have received any form of anti-tumor treatment previously.
2. Patients with allergic constitution and congenital immune deficiencies.
3. Patients who have undergone organ transplantation.
4. Patients with a history of severe bleeding tendencies or coagulation dysfunction; those who have had clinically significant bleeding symptoms within 1 month prior to the study treatment, including but not limited to gastrointestinal bleeding, hemoptysis; those who have received prolonged anticoagulation treatment within 10 days prior to the study treatment.
5. Patients who have experienced arteriovenous thrombotic events within 6 months before the study treatment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
6. Patients with active autoimmune diseases or inflammatory diseases, or a history thereof, including inflammatory bowel disease (e.g., colitis or Crohn's disease), diverticulitis (excluding diverticulosis), systemic lupus erythematosus, sarcoidosis or Wegener's granulomatosis (e.g., granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis). Exceptions to this criterion include patients with vitiligo or alopecia; patients with stable hypothyroidism after hormone replacement therapy (e.g., following Hashimoto's thyroiditis); patients with any chronic skin disease not requiring systemic treatment; inclusion of patients without active disease in the last 5 years is allowed only after consultation with the study physician.
7. Patients with active infections, including tuberculosis or human immunodeficiency virus (HIV 1/2 antibody positive).
8. Patients with uncontrollable complications, including but not limited to: persistent or active infections receiving study treatment (except HBV or HCV), symptomatic congestive heart failure, uncontrolled diabetes, uncontrolled hypertension, unstable angina, uncontrolled arrhythmias, active interstitial lung disease, severe chronic gastrointestinal disease with diarrhea, or any psychiatric/social situations that might limit compliance with study requirements, significantly increase the risk of adverse events (AE), or impair the ability of the patient to give written informed consent.
9. Pregnant or breastfeeding women.
10. Patients who do not agree to use effective contraception during the treatment period and for 3 months thereafter.
11. Patients participating in other clinical studies simultaneously.
12. Patients who are critically ill and unable to complete the investigation.
13. Patients with a history of other primary malignant tumors, except for the following: Malignant tumors treated with curative intent and no known active disease for ≥5 years prior to study treatment and with a low risk of relapse; adequately treated non-melanoma skin cancer or in-situ melanoma without evidence of disease; adequately treated carcinoma in situ without evidence of disease.
14. Patients with a history of psychiatric illness (e.g., schizophrenia, mania, anxiety disorder, depression, phobia) or diagnosed with a psychiatric disease at the time of enrollment or their spouses.
15. Patients or their spouses with communication barriers due to confusion, aphasia, intellectual disability, or other reasons that prevent normal responses.
16. Patients with other malignant neoplastic diseases.
17. Patients whom the researcher considers unsuitable for inclusion or whose participation might affect their ability to participate or complete the study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
pCR | After surgery (approximately 9-10 weeks after start of study treatment)
  Pathological complete response rate

SECONDARY OUTCOMES:
MPR | After surgery (approximately 9-10 weeks after start of study treatment)
  major pathological remission

OTHER OUTCOMES:
ORR | 9-10 weeks
  objective response rate
EFS | 1 years
  event free survival
OS | 2 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China